CLINICAL TRIAL: NCT00451035
Title: A Phase II, Multicentre Study of Oral LBH589 in Patients With Chronic Phase Chronic Myeloid Leukemia With Resistant Disease Following Treatment With at Least Two Fusion Gene of the BCR and ABL Genes (BCR-ABL) Tyrosine Kinase Inhibitors
Brief Title: Efficacy and Safety of LBH589 in Adult Patients With Refractory Chronic Myeloid Leukemia (CML) in Chronic Phase
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589B2202
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Results first posted 2021-07-14 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Chronic Myeloid Leukemia in Chronic Phase
Keywords: Refractory Chronic Myeloid Leukemia in Chronic Phase; adults; oral LBH589
MeSH Terms: interventions — Panobinostat

ARMS (1):
- Panobinostat (LBH589) (Experimental): Participants were administered panobinostat 20 milligram (mg) orally once a day (OD) three times a week as part of a 4 week (28 day) treatment cycle. Panobinostat were administered at the same time each morning with 8oz/240 milliliter (ml) of water after a fasting period of at least two hours (water was allowed). Participants could continue treatment until they experienced unacceptable toxicity or disease progression.
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589
  Other Names: Panobinostat

SUMMARY:
This study will evaluate the efficacy and safety of LBH589B in adult patients with chronic phase chronic myeloid leukemia with resistant disease following treatment with at least two BCR-ABL tyrosine kinase inhibitors

ELIGIBILITY:
Inclusion criteria:

* Male or female patients aged ≥ 18 years old
* Diagnosis of Philadelphia chromosome positive, chronic phase chronic myeloid leukemia
* Prior treatment with at least two BCR-ABL tyrosine kinase inhibitors with demonstrated resistance to the most recent kinase inhibitor therapy.
* Patients with a history of intolerance to one BCR-ABL kinase inhibitors will be considered eligible to enter the study if they demonstrate resistance to their most recent BCR-ABL kinase inhibitor.
* Patients who are intolerant of at least 2 BCR-ABL kinase inhibitors will be considered eligible to enter this study if they also demonstrate resistance to or intolerance of interferon-alpha (IFN-α) by the same criteria defined above.
* Patients must have adequate laboratory values:

  1. Hematology: absolute neutrophil count (ANC) ≥ 1.5 x 109/L, hemoglobin ≥ 8.0 g/dL.
  2. Serum chemistry: albumin ≥ 3 g/dL; aspartate aminotransferase (AST/GOT) and alanine aminotransferase (ALT/GPT) ≤ 2.5 x upper limit of normal (ULN) or ≤ 5.0 x ULN if the transaminase elevation is due to leukemic involvement; bilirubin ≤ 1.5 x ULN; creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥ 50 mL/min; potassium, phosphorus, magnesium and total calcium (corrected for serum albumin) or serum ionized calcium ≥ lower limit of normal (LLN), thyroid stimulating hormone (TSH) and free T4 (thyroxine) within normal limits.

Note: Potassium, calcium, and magnesium supplements to correct values that are < LLN, were allowed when documented as corrected prior to enrollment.

* Baseline measurement of left ventricular ejection fraction [assessment of the hearts ability to pump effectively]
* Assessment of patients ability to perform every day activities. Assessment by the Eastern Cooperative Oncology Group (ECOG) Performance Status

Exclusion criteria:

* A candidate for hematopoietic stem cell transplantation
* Prior therapy with certain medications
* Patients with a prior history of accelerated phase or blast crisis CML
* Impaired cardiac function or clinically significant cardiac diseases
* Concomitant use of certain medications. Therapeutic doses of sodium warfarin or any other anti-vitamin K drug (low doses for line patency were allowed). Prior HDACi treatment of CML, concomitant use of drugs with a risk of causing QT interval (QTc) prolongation or torsades de pointes, CYP3A4/5 inhibitors, anti-cancer therapy or radiation therapy, valproic acid (within 5 days prior to study drug treatment or during the study), chemotherapy or major surgery (within 3 weeks), immunotherapy (within 1 week), BCR-ABL tyrosine kinase inhibitors (TKI) ≤ 1 week of first treatment with panobinostat
* Impairment of GI function or GI disease
* Patients with unresolved diarrhea
* Patients who have received chemotherapy, any investigational drugs or undergone major surgery < 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who have received a BCR-ABL tyrosine-kinase inhibitor within 1 week of first treatment with LBH589
* Women who are pregnant or breast feeding or women of childbearing potential not using an effective method of birth control
* Male patients whose sexual partners are women of child bearing potential not using effective birth control

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-02-19 (Actual); Primary Completion 2008-04-13 (Actual); Study Completion 2008-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticlas, Study Director — Novartis Pharmaceuticals
Locations (10):
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Godinne
  - Novartis Investigative Site, Leuven
- Germany (7):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Munich

REFERENCES:
- [Result] Savelieva M, Woo MM, Schran H, Mu S, Nedelman J, Capdeville R. Population pharmacokinetics of intravenous and oral panobinostat in patients with hematologic and solid tumors. Eur J Clin Pharmacol. 2015 Jun;71(6):663-672. doi: 10.1007/s00228-015-1846-7. Epub 2015 May 5. PMID 25939707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 19 centers in multiple countries.
Pre-assignment Details: A total of 29 participants were enrolled, of which 29 participants discontinued the study treatment and 17 participants discontinued the study.
Groups:
- Panobinostat (LBH589): Participants were administered panobinostat 20 milligram (mg) orally once a day (OD) three times a week as part of a 4 week (28 day) treatment cycle. Panobinostat were administered at the same time each morning with 240 milliliter (ml) of water after a fasting period of at least two hours (water was allowed). Participants could continue treatment until they experienced unacceptable toxicity or disease progression.
Period: Overall Study
Arm/Group | Panobinostat (LBH589)
Started | 29
Completed | 12
Not Completed | 17
Not completed — Disease progression | 11
Not completed — Death | 3
Not completed — New anti-neoplastic therapy | 3

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all enrolled participants who have received at least one dose of study medication.
Groups:
- Panobinostat (LBH589): Participants were administered panobinostat 20 mg orally OD three times a week as part of a 4 week (28 day) treatment cycle. Panobinostat were administered at the same time each morning with 240 ml of water after a fasting period of at least two hours (water was allowed). Participants could continue treatment until they experienced unacceptable toxicity or disease progression.
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (12.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 26
  Black | 2
  Asian | 1

OUTCOME MEASURES:

1. Primary Outcome: Major (Complete/Partial) Cytogenetic Response (MCyR) Rate
Description: The CyR, based on the percentage of Ph+ metaphases by karyotype analysis on a bone marrow aspirate, was ideally assessed from a minimum of 20 metaphases in each bone marrow sample. The CyR was defined as: major response including complete (CCyR; 0% Ph+ metaphases) or partial (PCyR; 1 to 35% Ph+ metaphases), minor (36 to 65% Ph+ metaphases), minimal (66 to 95% Ph+ metaphases) or none (96 to 100% Ph+ metaphases).
Time Frame: From Start of the Study up to End of Study (approximately up to 19 Months)
Population: Full Analysis Set (FAS) consisted of all enrolled participants who have received at least one dose of study medication. The outcome measure was not achieved as the study was terminated due to insufficient clinical efficacy in the targeted participants population. Due to insufficient data, this outcome could not be measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 29
Participants | 0

2. Secondary Outcome: Duration of Major (Complete/Partial) Cytogenetic Response (MCyR) Rate
Description: The duration of response was defined as the time between the first documented response to the date of discontinuation due to progressive disease (PD) or death.
Time Frame: From Start of the Study up to End of Study (approximately up to 19 Months)
Population: The FAS consisted of all enrolled participants who have received at least one dose of study medication. The outcome measure was not achieved as the study was terminated due to insufficient clinical efficacy in the targeted participants population. Due to insufficient data, this outcome could not be measured.
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 0

3. Secondary Outcome: Complete Hematologic Response (CHR) Rate
Description: CHR was defined by meeting all criteria: white blood cell count < 10 x 109/L, platelet count < 450 x 109/L, myelocytes and metamyelocytes in peripheral blood < 5%, basophils in peripheral blood ≤ 5%, no myeloblasts or promyelocytes in peripheral blood, and no evidence of extramedullary involvement.
Time Frame: From Start of the Study up to End of Study (approximately up to 19 Months)
Population: as for outcome 2
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 0

4. Secondary Outcome: Complete Cytogenetic Response (CCyR) and Overall (Complete/Partial/Minor/Minimal) Cytogenetic Response (OCyR) Rates
Description: Cytogenetic response was assessed by bone marrow assessment based on the percentage of Ph+ metaphases by karyotype analysis on a bone marrow aspirate, was ideally assessed from a minimum of 20 metaphases in each bone marrow sample.
Time Frame: From Start of the Study up to End of Study (approximately up to 19 Months)
Population: as for outcome 2
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 0

5. Secondary Outcome: Major (MMR) and Complete (CMR) Molecular Response Rates
Description: Molecular response was defined as major (≤ 0.1% on the International Scale) and complete [absence of fusion gene of the BCR and ABL genes (BCR-ABL) on an quantitative reverse transcription polymerase chain reaction (qRT-PCR) assay with a sensitivity of at least 4.5 logs below baseline].
Time Frame: From Start of the Study up to End of Study (approximately up to 19 Months)
Population: as for outcome 2
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 0

6. Secondary Outcome: BCR-ABL Mutations of Participants at Study Entry and, in Responding Participants and at the Time of Disease Progression
Description: BCR-ABL messenger ribose nucleic acid (mRNA) expression (molecular response) was performed by quantitative polymerase chain reaction (qPCR) and mutational analysis was performed by direct sequencing technology, and both analyses were performed by Genzyme.
Time Frame: From Start of the Study up to End of Study (approximately up to 19 Months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 19
Participants | 0

7. Secondary Outcome: Progression Free Survival Time
Description: Progression-free survival time is defined as the time from the treatment start to the first documentation of the disease progression or the date of death, whichever occurs first
Time Frame: From Start of the Study up to End of Study (approximately up to 19 Months)
Population: as for outcome 2
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 0

8. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Panobinostat
Description: Cmax is defined as the Maximum (peak) plasma drug concentration after single dose administration. Cmax will be reported in units of nanogram/milliliter (ng/ML).
Time Frame: Pre-dose, and 0.25, 1-2, 3-4, 24, and 48 hours post-dose on Day 1
Population: The analysis was performed on Pharmacokinetic (PK) population, defined as all participants who provide at least one post-dose PK plasma sample. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 16
ng/mL | 9.1 (4.01)

9. Secondary Outcome: Time to Peak Concentration (Tmax) of Panobinostat
Description: Time to reach peak or maximum plasma drug concentration following drug administration. Tmax will be reported in units of hour (hr).
Time Frame: Pre-dose, and 0.25, 1-2, 3-4, 24, and 48 hours post-dose on Day 1
Population: The analysis was performed on PK population, defined as all participants who provide at least one post-dose PK plasma sample. Here, number of participants analyzed refer to the number of participants evaluable for this outcome at specified time point.
Measure: Median (Full Range); unit: hr
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 16
hr | 1.5 [0.2 to 3.6]

10. Secondary Outcome: Area Under the Plasma Concentration (AUC0-24) of Panobinostat
Description: Area under the curve (AUC) is defined as the area under concentration-time curve as a measure of drug exposure. The area under the plasma concentration-time curve from time zero to 24 hours.
Time Frame: Pre-dose, and 0.25, 1-2, 3-4, 24, and 48 hours post-dose on Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 12
ng*hr/mL | 96.0 (41.37)

11. Secondary Outcome: Last Observed Plasma Concentration (Clast) of Panobinostat
Description: Clast is defined as the Last observed (quantifiable) plasma concentration at last sampling time.
Time Frame: Pre-dose, and 0.25, 1-2, 3-4, 24, and 48 hours post-dose on Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 19
ng/mL | 1.8 (2.02)

12. Secondary Outcome: Time of Clast (Tlast) of Panobinostat
Description: Time of last sampling point. Tlast will be reported in units of hr
Time Frame: Pre-dose, and 0.25, 1-2, 3-4, 24, and 48 hours post-dose on Day 1
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 19
hr | 24.7 (16.19)

13. Secondary Outcome: QT Interval (QTc) in Participants Receiving Oral Panobinostat at Baseline and Change From Baseline to Extreme Value
Description: QTc monitoring was performed on specified days (Cycle1: Day1, 5 and 26), as well as a single pre-dose ECG once weekly during Cycle1: Week2 and Week3, Cycle2, and all subsequent cycles. Patient eligibility was ensured by a screening QTcF interval calculated by eResearchTechnology(eRT) prior to the baseline assessments. Treatment decisions were based on QTc determined by the automated reading at the investigational site (commonly used the Bazett's correction,QTcB) or measured and calculated by trained personnel at the site. Dosing relied on the investigator's assessment of the 6 baseline ECGs (the average of the 6pre-dose QTc intervals) performed prior to Cycle1/Day1 dosing, of the 3pre-dose ECGs during Cycle1:Day5 and 26, and of the single pre-dose ECGs performed once weekly for the remaining weeks of Cycle1 and subsequent cycles. The Baseline and Change From Baseline to Extreme Value QTcF interval for analysis was calculated by eRT based on the 6 baseline ECGs obtained on Cycle1/Day1.
Time Frame: From Start of the Study up to End of Study (approximately up to 19 Months)
Population: The analysis was performed on Safety population consisted of all participants who had received at least one dose of study medication and had one valid post-baseline assessment.
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Panobinostat (LBH589): Participants were administered panobinostat 20 mg orally OD three times a week as part of a 4 week (28 day) treatment cycle. Treatment were administered at the same time each morning with 240 milliliter (ml) of water after a fasting period of at least two hours (water was allowed). Participants could continue treatment until they experienced unacceptable toxicity or disease progression.
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 29
ms
  Baseline | 403.1 (23.45)
  Change from Baseline | 29.1 (23.91)

14. Secondary Outcome: Safety and Tolerability Profile of Oral Panobinostat
Description: Adverse events (AEs) are defined as any unfavorable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events (SAEs) are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.
Time Frame: From Start of the Study up to 28 Days After the last dose of Study Drug (approximately up to 19 Months)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Panobinostat (LBH589)
Number analyzed (Participants) | 29
Participants
  AEs | 28
  SAEs | 4
  Deaths | 3
  AEs leading to discontinuation | 6

ADVERSE EVENTS:
Time Frame: From Start of the Study up to 28 Days After the last dose of Study Drug (approximately up to 19 Months).
Description: Safety population consisted of all patients who received at least one dose of study medication and had one valid post-baseline assessment.
Groups:
- Panobinostat: Participants were administered panobinostat 20 mg orally OD three times a week as part of a 4 week (28 day) treatment cycle. Treatment were administered at the same time each morning with 240 ml of water after a fasting period of at least two hours (water was allowed). Participants could continue treatment until they experienced unacceptable toxicity or disease progression.
Arm/Group | Panobinostat
All-Cause Mortality (participants affected / at risk) | 3/29
Serious Adverse Events (participants affected / at risk) | 4/29
Other Adverse Events (participants affected / at risk) | 26/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat (N=29)
Leukocytosis (Blood and lymphatic system disorders) | 1
Splenic infarction (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panobinostat (N=29)
Anaemia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 3
Chills (General disorders) | 2
Fatigue (General disorders) | 8
Oedema peripheral (General disorders) | 5
Pyrexia (General disorders) | 5
Nasopharyngitis (Infections and infestations) | 2
White blood cell count increased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No